CLINICAL TRIAL: NCT06957951
Title: Effectiveness of WBV-Supported Core Training on Pain, Function, and Sleep in Lumbar Disc Herniation: A Randomized Controlled Trial
Brief Title: Effectiveness of WBV-Supported Core Training on Lumbar Disc Herniation
Acronym: WBV-LDH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Erzurum Technical University (Other); Ataturk University (Other)
Responsible Party: Principal Investigator, Esedullah Akaras, Dr., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETU-WBV-LDH-2023
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Lumbar Disc Herniation; Low Back Pain
Keywords: Whole-Body Vibration; Core Stabilization Exercises; Low Back Pain; Sleep Quality; Functional Disability
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physiotherapy (Active Comparator): Conventional Physiotherapy including hot pack, TENS, ultrasound, and education.
  Interventions: Other: Conventional Physiotherapy
- Core Stabilization Exercises (Active Comparator): Core stabilization exercises added to conventional physiotherapy.
  Interventions: Other: Conventional Physiotherapy; Behavioral: Core Stabilization Exercises
- WBV-Supported Core Exercises (Experimental): Participants received conventional physiotherapy combined with core stabilization exercises performed on a whole-body vibration platform (30 Hz, low amplitude ~2 mm).
  Interventions: Other: Conventional Physiotherapy; Behavioral: WBV-Supported Core Exercises

INTERVENTIONS:
Other: Conventional Physiotherapy — Application of hot packs, TENS (transcutaneous electrical nerve stimulation), therapeutic ultrasound, and posture/activity education for low back pain management.
Behavioral: Core Stabilization Exercises — Supervised core stabilization exercises including planks, bird-dog, and pelvic bridging, targeting trunk muscle strength and stability.
  Arms: Core Stabilization Exercises
Behavioral: WBV-Supported Core Exercises — Core stabilization exercises performed on a whole-body vibration platform (30 Hz frequency, low amplitude ~2 mm) during exercise execution to enhance neuromuscular stimulation.
  Arms: WBV-Supported Core Exercises

SUMMARY:
"This randomized controlled trial investigated the effects of conventional physiotherapy, core stabilization exercises, and WBV-supported core stabilization exercises on pain intensity, functional disability, quality of life, and sleep quality in male patients with lumbar disc herniation without neurological deficits."

DETAILED DESCRIPTION:
"This study aimed to compare the effects of whole-body vibration (WBV)-supported core exercises, standard core exercises, and conventional physiotherapy on pain, disability, quality of life, and sleep quality among male patients aged 30-50 years with lumbar disc herniation without neurological deficits. Participants were randomly allocated to one of three groups and underwent 12 sessions over 4 weeks. The outcomes assessed were pain (VAS), disability (ODI), quality of life (SF-36), and sleep quality (PSQI)."

ELIGIBILITY:
Inclusion Criteria:

* • Male gender

  * Age between 30 and 50 years
  * Diagnosis of lumbar disc herniation (L4-L5 or L5-S1)
  * No neurological deficits

Exclusion Criteria:

* • Prior lumbar surgery

  * Severe cardiopulmonary or musculoskeletal disorders
  * Uncontrolled systemic diseases
  * Participation in another clinical trial

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (VAS) | 4 weeks
  Change in pain scores measured by Visual Analog Scale.
Functional Disability (ODI) | 4 weeks
  Change in disability scores measured by Oswestry Disability Index.
Quality of Life (SF-36) | 4 weeks
  Change in quality of life scores
Sleep Quality (PSQI) | 4 weeks
  Change in sleep quality scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University Medical Faculty Physical Medicine and Rehabilitation Unit, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No